CLINICAL TRIAL: NCT01850212
Title: A Phase 4 Cross-Sectional Study of Bone Mineral Density in HIV-1 Infected Subjects
Status: Completed | Type: Observational
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Other Study IDs: GS-US-104-0423; 2011-004420-35 (EudraCT Number)
Record Dates: First submitted 2013-03-28; First posted 2013-05-09 (Estimated); Last update posted 2014-10-31 (Estimated); Status verified 2014-10

CONDITIONS: HIV Infections
Keywords: Treatment Experienced; Male greater than or equal to 50 years; Female postmenopausal
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- Male (≥ 50 years), TDF: Male (≥ 50 years of age) on regimens containing tenofovir disoproxil fumarate (TDF)
- Male (≥ 50 years of age), Non-TDF: Male (≥ 50 years of age) on non-TDF (tenofovir disoproxil fumarate) based nucleoside reverse transcriptase inhibitors (NRTIs)
- Female (Postmenopausal), TDF: Female (postmenopausal) on regimens containing tenofovir disoproxil fumarate (TDF)
- Female (Postmenopausal), Non-TDF: Female (postmenopausal) on non-TDF (tenofovir disoproxil fumarate) based NRTIs

SUMMARY:
A Phase 4 study is to characterize the profile of low bone mineral density (BMD) in ≥ 50 year old male subjects and post-menopausal female subjects on any tenofovir disoproxil fumarate (TDF)-based regimen

ELIGIBILITY:
Inclusion Criteria:

* Must have the ability to understand and sign a written informed consent form, which must be obtained prior to initiation of any study procedures.
* HIV-1 infected subjects regardless of race or ethnicity
* Use of one of the following taken as a stable, continuous, NRTI-containing antiretroviral (ARV) regimen for ≥ 3 years are allowed (within-class change of agents other than TDF within 3 years of study entry are permitted as specified):

  * TDF plus PI/r-containing regimen including subjects who switched from one TDF plus PI/r regimen to another TDF plus PI/r regimen
  * a TDF plus non-PI/r-containing regimen including subjects who switched from one TDF plus non-PI/r regimen to another TDF plus non-PI/r regimen
  * a Non-TDF NRTI plus a PI/r-containing regimen including subjects who switched from one non-TDF NRTI plus PI/r regimen to another non-TDF NRTI regimen plus PI/r regimen
  * a Non-TDF NRTI plus a non-PI/r-containing regimen including subjects who switched from one non-TDF NRTI plus non-PI/r regimen to another non-TDF NRTI regimen plus non-PI/r regimen
* Of note, subjects in the non-TDF groups must have never taken a regimen that includes TDF (including previous exposure to TDF for pre-exposure prophylaxis (PrEP))
* Subjects included in the TDF groups must have always taken a regimen that includes TDF. Non-PI/r agents include non-nucleoside reverse transcriptase inhibitors (NNRTIs), integrase inhibitors, triple nucleoside inhibitors and non-boosted protease inhibitors
* Male subjects must be ≥ 50 years of age
* Female subjects must be postmenopausal. Menopause can be assumed to have occurred in a woman when there is either appropriate medical documentation of prior complete bilateral oophorectomy or permanent cessation of previously occurring menses > 12 months as a result of ovarian failure or bilateral oophorectomy with documentation of hormonal deficiency by a certified healthcare provided
* Adequate records available to evaluate medical history for the 3 years prior to study entry

Exclusion Criteria:

* Subject has a contraindication to dual-energy X-ray absorptiometry (DEXA) scans
* Subject has a history of osteoporosis before initiating Highly Active Antiretroviral Treatment (HAART)

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Study population of ≥ 50 year old male subjects and post-menopausal female subjects
Sampling Method: Probability Sample
Enrollment: 476 (Actual)
Dates: Start 2013-02; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Femoral Neck and Spine (L1-4) T-score | Day 1
  Femoral neck and spine (L1-4) T-score will be used to characterize the profile of low bone mineral density (BMD) in ≥ 50 year old male subjects and post-menopausal female subjects on any tenofovir disoproxil fumarate (TDF)-based regimen relative to those on any non-TDF-based regimen for HIV infection.

SECONDARY OUTCOMES:
Observed T-score < -2 (yes/no) for femoral neck and spine (L1-4) | Day 1
  Observed T-score for femoral neck and spine will be used to further characterize low BMD.
Observed -2 ≤ T-score < -1 (yes/no) for femoral neck and spine (L1-4) | Day 1
  Observed T-score for femoral neck and spine will be used to further characterize low BMD.

CONTACTS AND LOCATIONS:
Overall Officials: Hiba Graham, Pharm D, Study Director — Gilead Sciences
Locations (73):
- Austria (5):
  - LKH Graz West, Graz
  - Medizinische Universitaet Innsbruck, Innsbruck
  - AKh Allgemeines Krankenhaus der Stadt Linz GmbH, Linz
  - Otto Wagner Spital, Vienna
  - Medizinische Universitat Wien, Vienna
- Belgium (5):
  - CHU Saint-Pierre University Hospital, Brussels
  - CUB Hopital Erasme- Free University of Brussels, Brussels
  - Cliniques Universitaires St. LUC (UCL), Brussels
  - UZ Leuven, Leuven
  - Centre Hospitalier Universitaire Sart Tilman Liège, Liège
- France (10):
  - Hôpital - Avicenne, Bobigny
  - Hôpital Saint André, Bordeaux
  - Groupe Hospitalier Pellegrin, Bordeaux
  - Hôpital Raymond Poincaré, Garches
  - Hôpital Croix-Rousse, Lyon
  - Maladie Infectieuses et Tropicales, Paris
  - Hôpital Cochin, Paris
  - Hopital Tenon, Paris
  - Hopital Haut-Leveque, Pessac
  - Centre Hospitalier de Tourcoing, Tourcoing
- Germany (14):
  - Gemeinschaftspaxis Dres. Jessen & Kollegen, Berlin
  - MVZ Ärzteforum Seestraße, Berlin
  - Charite-Universitatsmedizin Berlin, Berlin
  - MIB Dienstleistung GmbH, Berlin
  - Hopital Saint Antoine, Bonn
  - Universitatsklinik Koln (AöR), Cologne
  - Center for HIV and Hepatogastroenterology, Düsseldorf
  - Universitatsklinikum Erlangen, Erlangen
  - Universitäts-Hautklinik Essen, Essen
  - Klinikum der Johann Wolfgang Goethe Universitaet, Frankfurt
  - Infektionsmedizinisches Centrum Hamburg (ICH), Hamburg
  - Universitätskrankenhaus Eppendorf, Hamburg
  - MUC Research GmbH, München
  - Klinikum der Universität München-Großhadern, München
- UCD School of Medicine and Medical Sciences, Dublin, Ireland
- Italy (8):
  - Azienda Ospedaliero-Universitaria di Bologna - Policlinico S.Orsola-Malpighi, Bologna
  - Universitaria San Martino, Genova
  - Ospedale Luigi Sacco, Milan
  - Ospedale San Raffaele Turro, Milan
  - Azienda Ospedale San Paolo, Milan
  - Azienda Ospedaliero-Universitaria di Modena Policlinico, Modena
  - Ospedale Civile Spirito Santo, Pescara
  - Istituto Nazionale per le Malattie Infettive, Rome
- Netherlands (2):
  - Erasmus MC, Rotterdam
  - University Medical Center Utrecht, Utrecht
- Wroclawskie Centrum Zdrowia SP ZOZ, Wroclaw, Poland
- Portugal (5):
  - HPP Hospital de Cascais Dr. José de Almeida, Alcabideche
  - Hospital Santo António Capuchos, Lisbon
  - Hospital de Santa Maria, Lisbon
  - Hospital de Sao Joao, E.P.E., Porto
  - Hospital Joaquim Urbano, Porto
- Spain (6):
  - Hospital Germans Trias i Pujol, Badalona
  - Hospital Vall D'Hebron, Barcelona
  - Hospital Donostia, Donostia / San Sebastian
  - Hospital Ramón y Cajal, Madrid
  - Hospital Universitario La Paz, Madrid
  - Hospital Universitario Virgen del Rocio, Seville
- Sweden (2):
  - Sahlgrenska University Hospital - Dpt of Infectious Diseases, SU/Östra, Gothenburg
  - Karolinska University Hospital - Dept of Infectious Diseases, Stockholm
- Switzerland (2):
  - Universitätsklinik für Infektiologie, Bern
  - Cantons Hospital St. Gallen, Sankt Gallen
- United Kingdom (12):
  - Queen Elizabeth Hospital, Birmingham
  - Whittall Street Clinic, Birmingham
  - Birmingham Heartlands Hospital, Birmingham
  - Brighton & Sussex University Hospitals, Brighton
  - Royal London Hospital, London
  - Homerton University Hospital, London
  - Royal Free Hospital and University College London Hospital, London
  - Kings College London, London
  - Chelsea & Westminster Hospital, London
  - St. George's Hospital, London
  - Imperial College Healthcare NHS Trust St. Mary's Campus, London
  - Manchester Centre for Sexual Health, Manchester